CLINICAL TRIAL: NCT04910087
Title: Comparison of the Effect od Ketofol and Propofol on Intracranial Pressure Evaluated by Sonographic Optic Nerve Sheath Diameter Measurements in the Endoscopic Retrograde Cholangiopancreatography Procedures
Brief Title: The Effect of Anesthesia Management on Optic Nerve Sheath Diameter in the Ercp Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Anesthesiology Department, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: E1/1786/2021
Record Dates: First submitted 2021-05-26; First posted 2021-06-02 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Intracranial Pressure; Optic Nerve Sheath Diameter; Ketofol; Propofol
Keywords: Cholangiopancreatography, Endoscopic Retrograde; Intracranial Pressure; optic nerve sheath diameter; ketofol; propofol

STUDY DESIGN:
Intervention Model Description: Prospective randomized double blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group K: Ketofol (Active Comparator): A ketofol mixture of 15 cc propofol 2%, 2 cc ketamine 50 mg/ml, and 13 cc serum saline will be prepared in a 50 cc non-transparent syringe and delivered to the patient intravenously through perfuser device. (at a ratio of 100 mg ketamine/300 mg propofol) After the loading dose is administered at 1 mg/kg IV in 5 minutes based on propofol, 0.5 cc/kg/hour ketofol infusion will be initiated.
  If patients cannot tolerate the ERCP procedure or have a BIS value >85 or FPS (Faces Pain Scale)> 3, 0.25 mg/kg propofol will be administered as a separate IV push.
  Interventions: Diagnostic Test: Sonographic optic nerve sheath diameter measurement
- Group P: Propofol (Active Comparator): A propofol mixture of 15 cc propofol 2% and 15 cc serum saline will be prepared in a 50 cc non-transparent syringe and delivered to the patient intravenously through the perfuser device.
  After the loading dose is administered at 1 mg/kg IV propofol in 5 minutes ,0.5 cc/kg/hour propofol infusion will be initiated.
  If patients cannot tolerate the ERCP procedure or have a BIS value >85 or FPS (Faces Pain Scale)> 3, 0.25 mg/kg propofol will be administered as a separate IV push
  Interventions: Diagnostic Test: Sonographic optic nerve sheath diameter measurement

INTERVENTIONS:
Diagnostic Test: Sonographic optic nerve sheath diameter measurement — With the linear ultrasound probe operating at 11 MHz in B mode, it will be measured in 2 planes, 3.0 mm behind the optic disc, the transverse plane where the probe is placed horizontally and the sagittal plane where the probe is placed vertically. Then, the average of these measurements will be recorded for both eyes every 10 minutes.

SUMMARY:
Aim: To compare the effect of procedural anesthesia management with ketofol and propofol on the sonographic optic nerve sheath diameter in the endoscopic retrograde cholangiopancreatography (ERCP) procedures.

DETAILED DESCRIPTION:
Adequate visualization of the gastrointestinal mucosa during endoscopic retrograde cholangiopancreatography (ERCP) requires distention of the intestinal lumen by gas insufflation. High intraluminal pressures can increase intraabdominal pressure, leading to an increase in intracranial pressure. Ultrasonographic measurement of the optic nerve sheath diameter is a simple, non-invasive, and reliable technique for assessing intracranial pressure. Propofol, a sedative-hypnotic agent with rapid onset and short duration of action, is often used.Theoretically, the combination of ketamine and propofol may maintain sedation efficacy while reducing cardiovascular side effects through dose reduction and due to its synergistic effects.

The aim of this study is to demonstrate whether our anesthesia management has an effect on ICP change by measurement of optic nerve sheath diameter, predicting that insufflation performed for imaging during the ERCP procedure increase intraabdominal pressure, and frequently observed situations such as insufficient sedation, prone position, coughing and Valsalva during the procedure increase intracranial pressure (ICP).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ERCP procedure
* ASA score of I, II, and III

Exclusion Criteria:

* chronic lung disease
* renal or hepatic failure
* uncontrolled comorbidities (diabetes mellitus, hypertension, etc.)
* central nervous system disease
* pregnancy
* undergoing optic nerve surgery
* glaucoma or increased intraocular pressure, and retinal detachment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
optic nerve sheath diameter change among 6 time period | Baseline, immediately after anesthesia induction, immediately after gas insufflation, 10th minute of the ERCP procedure,20th minute of the ERCP procedure,immediately after completion of the ERCP procedure

CONTACTS AND LOCATIONS:
Overall Officials: ismail aytac, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No